CLINICAL TRIAL: NCT01583062
Title: Duration of Postoperative Antibiotic Prophylaxis in Facial Fractures (Mandibular Fractures, Zygomaticoorbital Fractures, Isolated Orbital Blow-out Fractures and LeFort I/II/III Fractures): 1 Day vs. 5 Days: a Prospective, Randomized, Double Blind and Placebo Controlled Study (Phase IV)
Brief Title: Duration of Postoperative Antibiotic Prophylaxis in Facial Fractures
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Limited number of patients
Sponsor: Insel Gruppe AG, University Hospital Bern (Other)
Collaborators: Schweizerische Unfallversicherung SUVA, Switzerland (Unknown); Mepha Parma AG, Switzerland (Unknown); GlaxoSmithKline AG, Switzerland (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 235/04; 1601 (Other: University Hospital Bern)
Record Dates: First submitted 2012-04-20; First posted 2012-04-23 (Estimated); Last update posted 2013-07-15 (Estimated); Status verified 2013-07

CONDITIONS: Surgical Wound Infection
Keywords: Surgical Wound Infection; Facial Injuries; Orbital Fractures; Zygomatic Fractures; Mandibular Fractures; Jaw Injuries
MeSH Terms: conditions — Surgical Wound Infection; Facial Injuries; Orbital Fractures; Zygomatic Fractures; Mandibular Fractures | interventions — Amoxicillin-Potassium Clavulanate Combination; Amoxicillin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Active Comparator): Both groups receive amoxicillin/clavulanic acid 1.2 g intravenously every eight hours from admission up to 24 hours postoperatively. Group 1 then receives amoxicillin/clavulanic acid 625 mg orally every eight hours for four days.
  Interventions: Drug: Amoxicillin/clavulanic acid
- 2 (Placebo Comparator): Both groups receive amoxicillin/clavulanic acid 1.2 g intravenously every eight hours from admission up to 24 hours postoperatively. Group 2 receives oral placebo using the same schedule for the same duration as group 1.
  Interventions: Drug: Amoxicillin plus placebo

INTERVENTIONS:
Drug: Amoxicillin/clavulanic acid — Both groups receive amoxicillin/clavulanic acid 1.2 g intravenously every eight hours from admission up to 24 hours postoperatively. Group 1 then receives amoxicillin/clavulanic acid 625 mg orally every eight hours for four days.
  Arms: 1
Drug: Amoxicillin plus placebo — Both groups receive amoxicillin/clavulanic acid 1.2 g intravenously every eight hours from admission up to 24 hours postoperatively. Group 2 receives oral placebo using the same schedule for the same duration as group 1.
  Arms: 2

SUMMARY:
Facial fractures make up a significant proportion of injuries in trauma patients. Treatment of these fractures often results in standard surgical interventions. While up to the early 1980's perioperative antibiotic prophylaxis in maxillofacial surgery was controversial, its efficacy is well accepted today. Chole and his team could show that the administration of antibiotics one hour preoperatively and eight hours after the intervention reduces the incidence of infectious complications in facial fractures from 42,2% to 8.9%. However there is still no consensus about the duration of the postoperative administration. In literature postoperative prophylaxis in facial fractures varies from single-shot 6-7 up to a duration of 7 and even ten days postoperatively 8-10. The use of antibiotics can be associated with allergic or toxic reactions, adverse effects, drug interactions and increasing bacterial resistance. In addition some authors assume that a prolonged administration of antibiotics might increase the risk of infectious complications via superinfection. On the other hand a short term or single shot administration might not be enough to prevent the onset of an postoperative infection. Up to date there is no standard to support the administration of antibiotics after surgical repair of a facial fracture.

The purpose of this prospective, randomized double-blinded trial is to investigate the utility of antibiotics administered in the postoperative period after surgical revision of facial fractures.

Hypothesis: a short-term antibiotic prophylaxis of 1 day postoperatively is equally effective as a long-term administration of 5 days in facial fractures.

DETAILED DESCRIPTION:
Background

While up to the early 1980's perioperative antibiotic prophylaxis in maxillofacial surgery was controversial its efficacy is well accepted today. Chole et al. showed that the administration of antibiotics reduces the incidence of infectious complications in facial fractures from 42,2% to 8.9%.

However there is still no consensus about the duration of the postoperative administration. In literature postoperative prophylaxis varies from single-shot up to 7 and even ten days postoperatively.

Antibiotic use is costly and associated with allergic reactions, toxic reactions, adverse effects, drug interactions and increasing bacterial resistance. Additionally some authors assume that a prolonged administration of antibiotics might even increase the risk of infectious complications via superinfection. On the other hand one might risk an increase of postoperative infections with a short term or single shot administration.

In a medline search only few studies could be found which deal with antimicrobial prophylaxis in maxillofacial surgery and in facial trauma surgery in particular.

Articles which advocate a single shot administration contain a very inhomogeneous group of patients. Merten et al. compared a single shot with a 48h regimen. The study included cleft patients, tumor resections, dental surgery, sinus revisions, plastic surgery and trauma. He concluded that a one shot administration of 1500mg cefuroxime is equally effective as a 48h regimen.

The second study which investigated the efficacy of single-dose antibiotic prophylaxis included preprosthetic, plastic, orthognathic, tumor and trauma surgery. Here also single shot administration was found to be sufficient in preventing postoperative infection. Studies about antibiotic single shot administration which included trauma patients only do not exist.

Some studies compared a 12 or 24 hour with a 5 day postoperative regime: Johnson et al. conducted a study with one hundred nine patients requiring pedicled flap reconstruction in the region of the head and neck. He investigated if 5 days of antibiotic administration would be more effective than 1 day and concluded that no beneficial effect from administration of antibiotics for longer than 24 hours postoperatively can be achieved in patients who undergo myocutaneous flap reconstruction.

Bentley et al. studied the effect on infection rates of 1-day and 5-day administration of prophylactic antibiotics in orthognathic surgical procedures. He concluded that antibiotic prophylaxis for orthognathic surgical procedures should continue beyond the immediate postoperative period for 5 days since the infection rate was significantly higher in the one day regimen (60% vs. 6.7%). It must be stated that in this study very strict criteria for wound infection (such as spontaneous wound dehiscence in the absence of pus drainage) were applied.

Abubaker et al. evaluated the difference between the effect of a 5-day postoperative course and a 12 hour administration of antibiotics in 30 Patients on the incidence of postoperative infection in uncomplicated fractures of the mandible. He concluded that a prolonged administration of antibiotics has no benefit in reducing the incidence of infections.

In other surgical fields guidelines concerning the perioperative antibiotic use have been established. The East practice management guidelines for example recommend to limit the postoperative administration in open fractures to 48 hours after wound closure. Unfortunately these guidelines can not be uncritically applied to maxillofacial trauma patients out of several reasons. Not only the fracture patterns are basically different from those in orthopedics but also the surgical treatment differs in many aspects: the impossibility of complete wound disinfection, the continuing contamination by saliva even after primary closure, the lack of casts or sterile wound dressings, the impossibility of extensive wound debridement or open wound treatment.

Pharmaceutical study substance:

Co-amoxiclav is an antibacterial combination consisting of the semisynthetic antibiotic amoxicillin and the ß-lactamase inhibitor, clavulanate potassium. It was introduced as "Augmentin®" in 1984 by Glaxosmithkline and Smithkline Beecham (collectively "GSK"). Since the patent expired in december 2002 several generic versions were approved.

It is used in the treatment of lower respiratory, middle ear, sinus, skin and urinary tract infections. In ENT and maxillofacial surgery it is used for prophylaxis and therapy for several indications. In the investigators' department the present prophylaxis regimen for facial fractures varies from 5 to 8 days postoperatively.

Objective

Aim of this study is to evaluate the difference between the effect of a five- vs. a one-day postoperative course of antibiotics on the incidence of postoperative infections in facial fractures.

Methods

Patients with a facial fractures, which need surgical revision, are randomly assigned into two groups. Both groups receive amoxicillin/clavulanic acid 1.2 g intravenously every eight hours from admission up to 24 hours postoperatively. Group A then receives amoxicillin/clavulanic acid 625 mg orally every eight hours for four days. Group B receives oral placebo using the same schedule for the same duration as group A. Follow up appointments are 1, 2, 4, 6 and 12 weeks and 6 months after surgery. The developement of a surgical site infection (according to CDC) is defined as primary end point.

ELIGIBILITY:
Inclusion Criteria:

* Isolated orbital fracture, zygomatic fracture, mandibular fracture, or LeFort I/II/III fracture which requires surgical treatment
* Written informed consent obtained

Exclusion Criteria

* Need of intensive care treatment
* Presence of an acute bacterial infection
* Gunshot wounds
* Pathological fracture
* Skull base fracture with rhinoliquorrhea or intracranial emphysema
* History of malignancy or radiation to the head and neck area
* Known hypersensitivity, allergy to penicillin or other beta-lactam antibiotics
* Reduced body weight (<40kg or BMI<17), severe renal insufficiency (stage 4 according to the Kidney Disease Outcomes Quality Initiative (KDOQI))
* Insufficient patient compliance

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 217 (Actual)
Dates: Start 2006-01; Primary Completion 2012-11 (Actual); Study Completion 2012-12 (Actual)

PRIMARY OUTCOMES:
Number of patients with infection | 6 months
  Infection according to Surgical site infection by CDC

SECONDARY OUTCOMES:
Number of patients with infection | 1 week
  Infection according to Surgical site infection by CDC
Number of patients with infection | 2 weeks
  Infection according to Surgical site infection by CDC
Number of patients with infection | 4 weeks
  Infection according to Surgical site infection by CDC
Number of patients with infection | 6 weeks
  Infection according to Surgical site infection by CDC
Number of patients with infection | 12 weeks
  Infection according to Surgical site infection by CDC
Number of days between trauma and first antibiotic administration | at dismissal from hospital, expected to be after 5 days
Number of days between trauma and operation | At dismissal from hospital, expected to be after 5 days
Location of fracture | At the end of surgery, expected to be after 90 minutes
Duration of surgery | At the end of surgery, expected to be after 90 minutes
  Measured in minutes
Number of patients with concomitant injuries | At the end of surgery, expected to be after 90 minutes

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Lieger, MD, DMD, Principal Investigator — Department of Oral and Maxillofacial Surgery, University Hospital Bern, Bern, Switzerland; Tateyuki Iizuka, MD, DDS, PhD, Study Chair — Department of Oral and Maxillofacial Surgery, University Hospital Bern, Bern, Switzerland
Locations (1):
- Dep. of Oral and Maxillofacial Surgery, Bern University Hospital, Bern, Switzerland

REFERENCES:
- [Background] Peterson LJ, Booth DF. Efficacy of antibiotic prophylaxis in intraoral orthognathic surgery. J Oral Surg. 1976 Dec;34(12):1088-91. PMID 1069110
- [Background] Martis C, Karabouta I. Infection after orthognathic surgery, with and without preventive antibiotics. Int J Oral Surg. 1984 Dec;13(6):490-4. doi: 10.1016/s0300-9785(84)80019-8. PMID 6439657
- [Background] Yrastorza JA. Indications for antibiotics in orthognathic surgery. J Oral Surg. 1976 Jun;34(6):514-6. PMID 1063838
- [Background] Chole RA, Yee J. Antibiotic prophylaxis for facial fractures. A prospective, randomized clinical trial. Arch Otolaryngol Head Neck Surg. 1987 Oct;113(10):1055-7. doi: 10.1001/archotol.1987.01860100033016. PMID 3304348
- [Background] Hotz G, Novotny-Lenhard J, Kinzig M, Soergel F. Single-dose antibiotic prophylaxis in maxillofacial surgery. Chemotherapy. 1994 Jan-Feb;40(1):65-9. doi: 10.1159/000239173. PMID 8306818
- [Background] Merten HA, Halling F. [Perioperative antibiotic prophylaxis in maxillofacial surgery]. Infection. 1993;21 Suppl 1:S45-8. doi: 10.1007/BF01710343. German. PMID 8314293
- [Background] Abubaker AO, Rollert MK. Postoperative antibiotic prophylaxis in mandibular fractures: A preliminary randomized, double-blind, and placebo-controlled clinical study. J Oral Maxillofac Surg. 2001 Dec;59(12):1415-9. doi: 10.1053/joms.2001.28272. PMID 11732026
- [Background] Folkestad L, Granstrom G. A prospective study of orbital fracture sequelae after change of surgical routines. J Oral Maxillofac Surg. 2003 Sep;61(9):1038-44. doi: 10.1016/s0278-2391(03)00316-1. PMID 12966479
- [Background] Gerlach KL, Pape HD. [Studies on preventive antibiotics in the surgical treatment of mandibular fractures]. Dtsch Z Mund Kiefer Gesichtschir. 1988 Nov-Dec;12(6):497-500. No abstract available. German. PMID 3253045
- [Background] National Kidney Foundation. K/DOQI clinical practice guidelines for chronic kidney disease: evaluation, classification, and stratification. Am J Kidney Dis. 2002 Feb;39(2 Suppl 1):S1-266. No abstract available. PMID 11904577
- See also: Click here for more information about the definition of Surgical Site Infections — http://www.cdc.gov/